CLINICAL TRIAL: NCT05369338
Title: The Effect of Low Level Light Therapy on Histamine- and Mucuna Pruriens-induced Pruritus in Healthy Volunteers: A Prospective, Double-blind, Randomised Sham-controlled Pilot Study
Brief Title: The Effect of Low Level Light Therapy on Histamine- and Mucuna Pruriens-induced Pruritus in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Kordula Lang-Illievich, MD, Medical University of Graz
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 33-431 ex 21/22
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomised, sham-controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subjects are blinded to the irradiation side by audiovisual masking (swimming goggles with blackened lenses, hearing protection). The subjects do not have access to the randomisation list and are not in the same room during the irradiation. This means that they are also blinded to the irradiation side.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Level Light Therapy (Experimental): The application of LLL is applied for 12 minutes using Repuls 7 (Repuls Lichtmedizintechnik GmbH, Vienna). This is a class IIb medical device. It applies pulsed red light of a frequency of 640nm. The intensity is 175 mWcm-2, which corresponds to a power density of 4,100 mW. The pulse frequency is set to 2.5 hz.
  The device is positioned 7cm from the skin using a distance ring.
  Interventions: Device: Low Level Light Therapy
- Sham controll (Sham Comparator): The application of LLL is applied for 12 minutes using Repuls 7 (Repuls Lichtmedizintechnik GmbH, Vienna). This is a class IIb medical device. It applies pulsed red light of a frequency of 640nm. The intensity is 175 mWcm-2, which corresponds to a power density of 4,100 mW. The pulse frequency is set to 2.5 hz.
  The device is positioned 7cm from the skin using a distance ring. The sham treatment is performed with the same device and the same distance ring without activating it.
  Interventions: Device: Sham Controll

INTERVENTIONS:
Device: Low Level Light Therapy — The application of LLL is applied for 12 minutes using Repuls 7 (Repuls Lichtmedizintechnik GmbH, Vienna). This is a class IIb medical device. It applies pulsed red light of a frequency of 640nm. The intensity is 175 mWcm-2, which corresponds to a power density of 4,100 mW. The pulse frequency is set to 2.5 hz.
  The device is positioned 7cm from the skin using a distance ring. The sham treatment is performed with the same device and the same distance ring without activating it.
  Other Names: LLLT
  Arms: Low Level Light Therapy
Device: Sham Controll — The application of LLL is applied for 12 minutes using Repuls 7 (Repuls Lichtmedizintechnik GmbH, Vienna). This is a class IIb medical device. It applies pulsed red light of a frequency of 640nm. The intensity is 175 mWcm-2, which corresponds to a power density of 4,100 mW. The pulse frequency is set to 2.5 hz.
  The device is positioned 7cm from the skin using a distance ring. The sham treatment is performed with the same device and the same distance ring without activating it.
  Arms: Sham controll

SUMMARY:
This is a prospective, double-blind, randomised, sham-controlled study whose primary aim is to test whether LLLT changes the intensity of itch after histamine application in healthy volunteers compared to sham application.

DETAILED DESCRIPTION:
Rationale and relevance of the study

Low-level light therapy (LLLT) is a method of photobiomodulation that involves the clinical application of light with wavelengths typically in the range of 600 to 1100 nm and with a typical power density of 5 mWcm² to 5 Wcm².

Clinical studies have demonstrated positive effects of LLLT on pain processing, which is attributed to a reduction in neurogenic inflammation and associated neuronal sensitisation. This has been proven by testing for hyperaesthesia or allodynia. In the course of neurogenic inflammation, histamine liberation also occurs, which can be associated with itching. Chronic itching is also frequently associated with somatosensory abnormalities in analogy to chronic pain. Itch-associated dysaesthesias, such as mechanical allocnesia and hyperknesia, can be seen as evidence of neuronal sensitisation in pruritus patients.

Oliviera et al. were able to demonstrate an antipruritic effect of LLLT in a case observation of five burn victims. By irradiating with laser, whose photobiomodulative mechanisms are similar to the mechanisms of LLL therapy, this effect was also investigated in lichen planus patients. The effect of LLL on pruritus can be demonstrated in the case observation of five burn victims.

Itch models can be divided into histamine-induced and non-histamine-induced. To date, there has been no structured investigation of the antipruritic effect of LLL, nor is it clear to what extent the itch-inducing mechanism has an influence on the suspected efficacy of LLL.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the participant
* Healthy test persons aged 18-60
* For female volunteers, negative pregnancy test

Exclusion Criteria:

* known allergy or hypersensitivity to histamine or the Mucuna pruriens
* history of skin diseases
* tattoos in the test area
* neoplasia in the test area
* pacemaker
* pregnancy
* epilepsy
* piercings
* fever
* local acute infection, skin inflammation/rashes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Pruritus Intensity | 2 minutes
  Histaminergic itch is determined using a visual analogue scale (0-100) The non-histaminergic itch is determined by means of a visual analogue scale (0-100).

SECONDARY OUTCOMES:
Neurogenic inflammation | 10 minutes
  The neurogenic inflammation of histaminergic itch is determined by recording the flare area and measuring the skin temperature.
  The neurogenic inflammation of non-histaminergic itch is determined by recording the flare area and measuring the skin temperature.
Alloknesia | 10 minutes
  an area of alloknesia will be tested in the histaminergic itch model using cotton swabs.
  an area of alloknesia is tested in the non-histaminergic itch model using cotton swabs.
Hyperknesia | 10 minutes
  a hyperkneesia area is tested in the histaminergic itch model using a von Frey filament.
  a hyperkneesia area is tested in the non-histaminergic itch model using a von Frey filament.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical university of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No